CLINICAL TRIAL: NCT05909098
Title: Xiangyang No.1 People's Hospital, Hubei University of Medicine
Brief Title: Safety and Efficacy of Autologous NK Cell Adjuvant Therapy for Relapsed/Refractory Non-Hodgkin's B-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangyang No.1 People's Hospital (Other)
Collaborators: Qingdao Haier Biotechnology Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Bin Pei, Director, Xiangyang No.1 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xiangyang1PH
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: NK Cell; B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cell (Experimental): autologous NK cell adjuvant therapy
  Interventions: Combination Product: autologous NK cell

INTERVENTIONS:
Combination Product: autologous NK cell — autologous NK cell

SUMMARY:
This study was a single-arm trial of autologous NK cell adjuvant therapy for relapsed/refractory non-Hodgkin's B-cell lymphoma. The locations isXiangyang No.1 People's Hospital, Hubei University of Medicine. The population was relapsed/refractory non-Hodgkin's B-cell lymphoma. The sample size was 33. The intervention was R-GemOx regimen combined with autologous NK cells. The dose of autologous NK cells was body surface area x (2-4) x 109 cells. The course of treatment was once every 14 days. The primary outcome measure was ORR. The duration of assessment was for each treatment cycle, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 3 years, and 5 years of treatment.

DETAILED DESCRIPTION:
This study was a single-arm trial of autologous NK cell adjuvant therapy for relapsed/refractory non-Hodgkin's B-cell lymphoma. The locations isXiangyang No.1 People's Hospital, Hubei University of Medicine. The population was relapsed/refractory non-Hodgkin's B-cell lymphoma. The sample size was 33. The intervention was R-GemOx regimen combined with autologous NK cells. The dose of autologous NK cells was body surface area x (2-4) x 109 cells. The course of treatment was once every 14 days. The primary outcome measure was ORR. The duration of assessment was for each treatment cycle, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 3 years, and 5 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age 15 years to 80 years, with life expectancy greater than 6 months.
2. Pathologically confirmed non-Hodgkin B-cell lymphoma, confirmed by pathological examination at a grade A class 3 hospital or above, with pathology reported less than 3 years ago.
3. First diagnosed relapsed/refractory non-Hodgkin's B-cell lymphoma.
4. ECOG scores were 0 to 2
5. Presence of at least one CT measurable lesion locus with a maximum transverse diameter of ≥1.5 cm before inclusion in the study.
6. For women of childbearing potential, a negative pregnancy test must be confirmed before inclusion in the study and no intention to have children within 2 years.
7. For men of childbearing potential, inform and require the use of an effective barrier contraceptive method.
8. Volunteer to participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Presence of bone marrow or/and central nervous system lymphoma.
2. Patients with less than 5% peripheral blood NK cell percentage and pre-culture failure.
3. Combined with other malignancies.
4. Fever of non-disease-related origin within the last 5 days.
5. Presence of uncontrollable bacterial, fungal, viral or other infections.
6. Patients with HIV, TP positive
7. Patients with severe cardiopulmonary, hepatic and renal, and cerebral dysfunction are present.
8. Presence of other serious diseases that conflict with this protocol, such as autoimmune diseases, immunodeficiencies, severe thrombocytopenia, platelet dysfunction syndrome, etc.
9. Received any form of organ transplantation, including allogeneic stem cell transplantation.
10. Presence of a serious psychiatric disorder.
11. Inability to communicate normally and incapacitation make it difficult to assess the safety and effectiveness of treatment.
12. Pregnant or lactating women.
13. The researchers deemed unsuitable for participation in this study. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard

SECONDARY OUTCOMES:
CR | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
PR | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
SD | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
PD | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
CBR | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
PFS | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
DOR | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
OS | up to 5 years of treatment
  Refer to the 2014 version of Lugano standard
ECOG | up to 5 years of treatment
  ECOG score Zubrod-ECOG-WHO (ZPS, 5-point scale)
EORTC QLQ-C30 | up to 5 years of treatment
  EORTC:The European O-rganization for Reasearch and Treatment of Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bin Pei, Principal Investigator — Xiangyang No.1 People's Hospital
Locations (1):
- EC of Xiangyang No.1 People's Hospital Hubei University of Medicine, Hubei, Xiangyang, China

IPD SHARING:
Plan to Share IPD: No